CLINICAL TRIAL: NCT04586036
Title: The Evaluation of Ankle Joint Braces Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Łysoń (Other)
Responsible Party: Sponsor-Investigator, Barbara Łysoń, master of science, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DS-295
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Ankle Injuries; Ankle Sprains
Keywords: ankle joint brace; atfl; oxford foot model
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- young healthy adults (Experimental): Gait measured by Vicon Nexus System
  Interventions: Other: ankle joint brace 1; Other: ankle joint brace 2; Other: ankle joint brace 3; Other: ankle joint brace 4; Other: ankle joint brace 5
- young adults with chronic ankle joint instability (Experimental): Gait measured by Vicon Nexus System
  Interventions: Other: ankle joint brace 1; Other: ankle joint brace 2; Other: ankle joint brace 3; Other: ankle joint brace 4; Other: ankle joint brace 5

INTERVENTIONS:
Other: ankle joint brace 1 — The influence of ankle joint brace 1 on gait biomechanics
Other: ankle joint brace 2 — The influence of ankle joint brace 2 on gait biomechanics
Other: ankle joint brace 3 — The influence of ankle joint brace 3 on gait biomechanics
Other: ankle joint brace 4 — The influence of ankle joint brace 4 on gait biomechanics
Other: ankle joint brace 5 — The influence of ankle joint brace 5 on gait biomechanics

SUMMARY:
The project concerns the evaluation of commercially available ankle joint braces effectiveness used as orthopedic supply after ankle joint ligaments tear injury. Authors hypothesize that the restriction of range of motion may be not sufficient in the early healing process.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35
* female or male
* good health condition
* chronic ankle joint instability (for chronic ankle instability group)

Exclusion Criteria:

* lower limb injuries (last 6 months)
* extreme sports athletes
* no chronic ankle joint instability (for chronic ankle instability group)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Oxford Foot Model Angles | 2 hours
  Ankle angles, Hindfoot Tibia angles and Forefoot Hindfoot angles caculated by Oxford Foot Model, colected with the use of Vicon Motion Capture system

CONTACTS AND LOCATIONS:
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Mazowsze, Poland